CLINICAL TRIAL: NCT00386971
Title: Effects of L-Carnitine on Postprandial Clearance of Triglyceride-rich Lipoproteins in HIV Patients on HAART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200614280; GCRC protocol 109
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Hyperlipidemia; HIV Infections
Keywords: L-carnitine; HIV; TGRL metabolism; postprandial; HIV Treatment Experienced
MeSH Terms: conditions — Hyperlipidemias; HIV Infections | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): L-carnitine
  Interventions: Dietary Supplement: L-carnitine
- 2 (Placebo Comparator): Placebo
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: L-carnitine — 3 grams daily in liquid form by mouth
  Arms: 1
Other: placebo — 1 oz sweet tasting liquid daily by mouth
  Arms: 2

SUMMARY:
Included in this study will be patients with HIV and being treated with highly active antiretroviral medications (HAART) including protease inhibitors (PI) or non-nucleoside reverse transcriptase inhibitors (NNRTI). Protease inhibitors and non-nucleoside reverse transcriptase inhibitors are very common medications in HIV treatment and are usually given with other medications as part of a standard treatment for HIV (HAART).

We hope to learn more about how the levels of cholesterol-and triglyceride-carrying particles (lipoproteins) are affected by a nutritional supplement, L-Carnitine, in HIV-positive patients treated with antiretroviral medications.

DETAILED DESCRIPTION:
The postprandial state is a proinflammatory and proatherogenic condition. Increasing evidence support the contention the elevated triglyceride (TG)-rich lipoproteins (TGRL) are atherogenic. Hypertriglyceridemia is a characteristic of the metabolic complications during human immunodeficiency virus/highly active antiretroviral therapy (HIV/HAART) and the increased postprandial lipemia commonly seen in this situation may convey an increased cardiovascular risk. A possible contribution to the hypertriglyceridemia in HIV/HAART may be a decrease in mitochondrial function, resulting in a decreased fatty acid oxidation. A decrease in mitochondrial function may also contribute to insulin resistance. L- Carnitine plays an important role in the transfer of long-chain acyl groups into the mitochondrial matrix and potentially improves energy metabolism. L- Carnitine has been shown to reduce hypertriglyceridemia during HAART in HIV-positive subjects, but virtually nothing is known about its effect in the postprandial state. We have experience from postprandial studies in HAART-treated HIV-positive African American and Hispanic subjects, where we have focused on the relationship between lipids, fatty acids, insulin and adipokines. This is of particular relevance among African Americans, where key metabolic components differ substantially from levels in Caucasians. Further, the relationship between metabolic parameters and HIV/HAART is far less explored in this ethnic group. We recently found a proportional relationship between insulin and non-esterified fatty acids (NEFA) in response to food among African American HIV-positive subjects. Further, we showed a relationship between fasting insulin and postprandial adipokine levels.

In this randomized, double blind placebo-controlled pilot study, we will explore whether L- Carnitine affects TGRL metabolism in the fasting and the postprandial states among African American and Hispanic HIV-positive subjects undergoing antiretroviral therapy.

We hypothesize: (1) that L- Carnitine supplementation will improve both fasting TGRL levels and the postprandial response, and (2) that L- Carnitine will impact on the relationship between insulin and NEFA or adipokines in the postprandial state.

In our specific aims, we will test the effect of L- Carnitine supplementation on:

* Baseline TGRL metabolism and insulin, NEFA and adipokine levels
* Postprandial TGRL responses and the postprandial relationship between insulin and non-esterified fatty acids (NEFA) and adipokines We believe that the results generated from the proposed studies will help to evaluate effects of L- Carnitine supplementation on postprandial TGRL-associated cardiovascular risks.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women Ages 18-70,
* Stable HAART regimen x 6 mo,
* PI or NNRTI based regimens,
* Caucasian, African American or Hispanic patients

Exclusion Criteria:

* Diabetes Mellitus,
* Liver Disease,uncontrolled
* Pregnant or nursing mothers,
* BMI> 35,
* Hemoglobin <11 g/dl,
* Conditions known to lower seizure threshold (ie. brain tumor) or taking medications that lower seizure threshold,
* Patients taking: Warfarin, ValproicAcid or Zidovudine,Wellbutrin or Effexor
* Chronic Kidney Disease Stage 3-5,
* Untreated Thyroid Disease,
* Hormone replacement therapy,
* Triglycerides >500 mg/dl (fasting)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
L-carnitine supplementation will improve fasting TGRL levels and the postprandial response | 6 weeks

SECONDARY OUTCOMES:
L-carnitine will impact upon the relationship between insulin and NEFA or adipokines in the postprandial state | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lars Berglund, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- GCRC UC Davis, Sacramento, California, United States